CLINICAL TRIAL: NCT05190289
Title: The Relationship Between Paraspinal Muscle Degeneration and Bone Mass and Clinical Outcomes After Surgery in Patients With Lumbar Degenerative Diseases
Brief Title: Paraspinal Muscle Degeneration, Bone Mass and Clinical Outcomes in Patients With Lumbar Degenerative Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021134
Record Dates: First submitted 2021-06-27; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-06

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Scoliosis
Keywords: Degenerative Lumbar Disease; Clinical Outcome; Complication; Paraspinal Muscle; Bone Mass
MeSH Terms: interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Compared Group: Patients without inferior clinical outcomes
  Interventions: Other: Pre-existing degenerative factors of paraspinal muscles and bone mass
- Case Group: Patients with inferior clinical outcomes
  Interventions: Other: Pre-existing degenerative factors of paraspinal muscles and bone mass

INTERVENTIONS:
Other: Pre-existing degenerative factors of paraspinal muscles and bone mass — Pre-existing degenerative factors of paraspinal muscles, including muscle atrophy and fat infiltration; bone mass

SUMMARY:
This study was a retrospective study. The investigators intended to review the preoperative paraspinal muscle imaging data of patients with lumbar spinal stenosis and degenerative scoliosis treated in hospital, and follow up the symptoms, quality of life and surgical complications at 1 year and at the last follow-up. The aims were: (1) to explore the correlation between paraspinal muscle imaging parameters and clinical outcomes; (2) based on the postoperative functional scores and the presence of complications, to explore the best combination of imaging parameters for predictive value of prognosis; (3) to evaluate the consistency between different measurement methods, and improve the standardized paraspinal muscle imaging assessment; (4) Combining the characteristics of individual bone mass and paravertebral muscle (functional and imaging assessment), to explore the correlation between bone loss and paravertebral muscle degeneration; (5) to explore a muscle-bone mass assessment system that could reflect the prognosis of patients.

DETAILED DESCRIPTION:
This study was a retrospective study. The investigators intended to review the preoperative paraspinal muscle imaging data of patients with lumbar spinal stenosis and degenerative scoliosis treated in our hospital, and follow up the symptoms, quality of life and surgical complications at 1 year and at the last follow-up. The aims were: (1) to explore the correlation between paraspinal muscle imaging parameters and clinical outcomes; (2) based on the postoperative functional scores and the presence of complications, to explore the best combination of imaging parameters for predictive value of prognosis; (3) to evaluate the consistency between different measurement methods, and improve the standardized paraspinal muscle imaging assessment; (4) Combining the characteristics of individual bone mass and paravertebral muscle (functional and imaging assessment), to explore the correlation between bone loss and paravertebral muscle degeneration; (5) to explore a muscle-bone mass assessment system that could reflect the prognosis of patients.

The investigators intended to review the patients who underwent posterior surgery for degenerative lumbar diseases from January 2010 to December 2019.

1. To review the patients who underwent posterior surgery in orthopedic department for degenerative scoliosis. The inclusion criteria were: (1) above the age of 45; (2) satisfy at least one of the following criteria: cobb angle > 10°, sagittal vertical axis (SVA) > 5cm, pelvic tilt (PT) > 25°, or thoracic kyphosis (TK) > 60°. The exclusion criteria were: (1) with a history of arthritic tumor or neuromuscular disease (2) with a history of spinal surgery.
2. To review the patients who underwent posterior surgery in orthopedic department for lumbar spinal stenosis. The inclusion criteria were: (1) above the age of 45; (2) diagnosis of lumbar spinal stenosis. The exclusion criteria were: (1) with a history of arthritic tumor or neuromuscular disease (2) with a history of spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Underwent posterior surgery for degenerative scoliosis;
* Above the age of 45;
* Satisfy at least one of the following criteria: cobb angle > 10°, sagittal vertical axis > 5cm, pelvic tilt > 25°, or thoracic kyphosis > 60°.

Exclusion Criteria:

* Underwent posterior surgery for lumbar spinal stenosis;
* Above the age of 45;
* Diagnosis of lumbar spinal stenosis.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In the orthopaedic department of Peking University Third Hospital, patients with a clear diagnosis of lumbar degenerative diseases, and were performed by posterior surgery will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-03 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Disability | 12 months; through study completion, an average of 3 years
  The Oswestry Disability Index (ODI) (0-100, high score indicates severer disability) is used to assess disability.
Low Back pain | 12 months; through study completion, an average of 3 years
  The Visual Analog Scale (VAS) (0-10, high score indicates more pain) is used to evaluate leg pain.
Leg pain | 12 months; through study completion, an average of 3 years
  The Visual Analog Scale (VAS) (0-10, high score indicates more pain) is used to evaluate leg pain.
Sagittal balance | 12 months; through study completion, an average of 3 years
  Sagittal balance is evaluated by anteroposterior and lateral X-ray of the whole spine at the standing position.
Bone nonunion | 12 months; through study completion, an average of 3 years
  Bone nonunion was evaluated by dynamic X-ray. Bone nonunion was defined as 1) there was no continued bone fusion mass at any fusion segment; 2) any motion (greater than 3 mm or 3°) on flexion/ extension plain radiographs.
Screw loosening | 12 months; through study completion, an average of 3 years
  Screw loosening was evaluated on spine radiograph or CT. Screw loosening was defined when a 1mm or wider circumferential radiolucent line around the pedicle screw was confirmed.
Proximal junctional kyphosis | 12 months; through study completion, an average of 3 years
  Proximal junctional angle (PJA) was determined by the sagittal angle subtended by the inferior endplate of the uppermost instrumented vertebra (UIV) and the superior end plate of the vertebrae two levels above the UIV (UIV + 2). The definition of proximal junctional kyphosis (PJK) was PJA 10 or greater and at least 10 greater than the corresponding preoperative measurement.
Proximal scoliosis progression | 12 months; through study completion, an average of 3 years
  The proximal scoliosis progression (PSP) was defined as the disc wedging increased 10 degrees from postoperative to two-year follow up on the AP radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Shi Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will make the clinical study report available for half a year after the publication of the results of the study.
Supporting Information: CSR
Time Frame: The individual participant data (IPD) will become available for half a year after the publication of the results of the study.
Access Criteria: The IPD is available to the readers of the journal in which our research is published. The corresponding author of the published papers will review the requests.

REFERENCES:
- [Result] Ropponen A, Videman T, Battie MC. The reliability of paraspinal muscles composition measurements using routine spine MRI and their association with back function. Man Ther. 2008 Aug;13(4):349-56. doi: 10.1016/j.math.2007.03.004. Epub 2007 Jun 6. PMID 17556006
- [Result] Anderson DE, Bean JF, Holt NE, Keel JC, Bouxsein ML. Computed tomography-based muscle attenuation and electrical impedance myography as indicators of trunk muscle strength independent of muscle size in older adults. Am J Phys Med Rehabil. 2014 Jul;93(7):553-61. doi: 10.1097/PHM.0000000000000059. PMID 24508931
- [Result] Cooley JR, Walker BF, M Ardakani E, Kjaer P, Jensen TS, Hebert JJ. Relationships between paraspinal muscle morphology and neurocompressive conditions of the lumbar spine: a systematic review with meta-analysis. BMC Musculoskelet Disord. 2018 Sep 27;19(1):351. doi: 10.1186/s12891-018-2266-5. PMID 30261870
- [Result] Crawford RJ, Cornwall J, Abbott R, Elliott JM. Manually defining regions of interest when quantifying paravertebral muscles fatty infiltration from axial magnetic resonance imaging: a proposed method for the lumbar spine with anatomical cross-reference. BMC Musculoskelet Disord. 2017 Jan 19;18(1):25. doi: 10.1186/s12891-016-1378-z. PMID 28103921
- [Result] Hong X, Shi R, Wang YT, Liu L, Bao JP, Wu XT. Lumbar disc herniation treated by microendoscopic discectomy : Prognostic predictors of long-term postoperative outcome. Orthopade. 2018 Dec;47(12):993-1002. doi: 10.1007/s00132-018-3624-6. PMID 30171289
- [Result] Zotti MGT, Boas FV, Clifton T, Piche M, Yoon WW, Freeman BJC. Does pre-operative magnetic resonance imaging of the lumbar multifidus muscle predict clinical outcomes following lumbar spinal decompression for symptomatic spinal stenosis? Eur Spine J. 2017 Oct;26(10):2589-2597. doi: 10.1007/s00586-017-4986-x. Epub 2017 Feb 8. PMID 28180981
- [Result] Storheim K, Berg L, Hellum C, Gjertsen O, Neckelmann G, Espeland A, Keller A; Norwegian Spine Study Group. Fat in the lumbar multifidus muscles - predictive value and change following disc prosthesis surgery and multidisciplinary rehabilitation in patients with chronic low back pain and degenerative disc: 2-year follow-up of a randomized trial. BMC Musculoskelet Disord. 2017 Apr 4;18(1):145. doi: 10.1186/s12891-017-1505-5. PMID 28376754
- [Result] Pennington Z, Cottrill E, Ahmed AK, Passias P, Protopsaltis T, Neuman B, Kebaish KM, Ehresman J, Westbroek EM, Goodwin ML, Sciubba DM. Paraspinal muscle size as an independent risk factor for proximal junctional kyphosis in patients undergoing thoracolumbar fusion. J Neurosurg Spine. 2019 May 31;31(3):380-388. doi: 10.3171/2019.3.SPINE19108. Print 2019 Sep 1. PMID 31151107
- [Result] Betz M, Burgstaller JM, Held U, Andreisek G, Steurer J, Porchet F, Farshad M; LSOS Study Group. Influence of Paravertebral Muscle Quality on Treatment Efficacy of Epidural Steroid Infiltration or Surgical Decompression in Lumbar Spinal Stenosis-Analysis of the Lumbar Spinal Outcome Study (LSOS) Data: A Swiss Prospective Multicenter Cohort Study. Spine (Phila Pa 1976). 2017 Dec 1;42(23):1792-1798. doi: 10.1097/BRS.0000000000002233. PMID 28542102